## BOSTON MEDICAL CENTER AND THE BOSTON UNIVERSITY SCHOOLS OF MEDICINE, PUBLIC HEALTH AND DENTAL MEDICINE





## NCT06455111

H-41743 PI Dr. Nicole Spartano

## CGM Interpretation without Diabetes Study RESEARCH INFORMATION SHEET

You are being asked to voluntarily participate in a research study. We are conducting this study to investigate concordance among endocrinologists in recommending follow-up measures based on continuous glucose monitor (CGM) reports for patients without diabetes. We are asking you to complete our survey because you are a clinician with expertise in CGM. If you agree, we will ask you to evaluate 20 CGM reports from deidentified research participants. Based on these reports, you will be asked whether you would classify the participant's results as warranting follow-up with a healthcare provider, not warranting follow-up, or reflecting a potential CGM error.

We will ask you to provide your name and email address if you would like to participate as an author on the publication of our survey results. Your name and email will be stored separately from your survey responses. Otherwise, we will not ask for your name. We will store electronic files in computer systems with password protection and encryption. However, we cannot guarantee complete confidentiality.

After you complete the survey, please email Nicole to let her know you would like to participate in the interpretation of our survey results as an author.

If you have any questions, please contact Nicole Spartano, PhD, spartano@bu.edu, 315-415-2040.